CLINICAL TRIAL: NCT01728610
Title: Effect of Probiotic Supplement in Alleviating Functional Gastrointestinal Symptoms (IBS-2)
Brief Title: Effect of Probiotic Supplement in Alleviating Functional Gastrointestinal Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Danisco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IBS-2
Record Dates: First submitted 2012-10-05; First posted 2012-11-20 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; probiotic; pain; bloating; diarrhoea; constipation
MeSH Terms: conditions — Irritable Bowel Syndrome; Pain; Diarrhea; Constipation | interventions — Probiotics; Lacteol; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active high (Active Comparator): Probiotic, high dose
  Interventions: Dietary Supplement: Probiotic (Active high)
- Active low (Active Comparator): Probiotic, low dose
  Interventions: Dietary Supplement: Probiotic (Active low)
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic (Active high) — Higher dose of probiotic supplement
  Other Names: Lactobacillus
  Arms: Active high
Dietary Supplement: Probiotic (Active low) — Lower dose of probiotic supplement
  Other Names: Lactobacillus
  Arms: Active low
Dietary Supplement: Placebo — Placebo
  Other Names: Maltodextrin as placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to analyse the effect of a probiotic supplement on functional intestinal symptoms among subjects diagnosed with irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
The aim of the intervention is to analyse the effect of a probiotic supplement in a dose-responsive set up on functional intestinal symptoms among subjects diagnosed with IBS according to Rome III criteria. Subjective assessment of bowel symptoms, quality of life, anxiety and depression and adequate relief will be assessed as with questionnaires as outcome measures. The intestinal microbiota will be analysed from faecal samples.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 65 fulfilling Rome III criteria for IBS will be recruited. Sufficient general health and orientation for participating in the study is required and will be evaluated by the MDs.

Exclusion Criteria:

* Diagnosed or suspected organic gastrointestinal diseases or severely impaired general health.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 391 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in functional bowel symptoms | 0 weeks, 4 weeks, 12 weeks
  Validated questionnaire

SECONDARY OUTCOMES:
Change in quality of life | 0 weeks, 4 weeks, 12 weeks
  Validated questionnaire
Change in anxiety and depression | 0 weeks, 4 weeks and 12 weeks
  Validated questionnaire
Adequate relief | Weekly over 3 month intervention
  Weekly question
Change in faecal microbiota | 0 weeks, 4 weeks, 12 weeks
  Detection and quantification of microbes from faecal samples
Safety of investigational product | Throughout the intervention phase
  Recording of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lea Veijola, MD, Principal Investigator — Herttoniemi Hospital; Arthur Ouwehand, PhD, Study Chair — DuPont Nutrition and Health; Sampo Lahtinen, PhD, Study Chair — DuPont Nutrition and Health; Anna Lyra, PhD, Study Director — DuPont Nutrition and Health
Locations (2):
- Finland (2):
  - Mehiläinen Töölö, Helsinki, Helsinki
  - Mehiläinen Turku, Turku, Turku

IPD SHARING:
Plan to Share IPD: No